CLINICAL TRIAL: NCT06227858
Title: Investigation of the Psychological and Physiological Effects of a Standardised Saffron Extract Supplementation on Symptoms Associated to Perimenopause in Healthy Older Women: A Randomised Double-blind, Placebo-Controlled, Parallel-group Clinical Trial
Brief Title: Effects of a Standardised Saffron Extract Supplementation on Symptoms Associated With Perimenopause in Healthy Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of East Anglia (Other); Activ'inside (Industry)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LUMHS/REC/-221
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Perimenopausal Disorder

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation will be processed by computer-generated random sequence number and will be performed by an independent member of the medical support team which will not be involved in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saffron extract supplementation (15mg, twice daily) (Experimental): The experimental group will take a single capsule containing: 15mg of of saffron extract (stigma of the flower Crocus sativus), 340mg of Maltodextrin, encapsulated in hydroxypropyl methyl cellulose (HPMC), twice daily (one morning and one evening after the meal).
  Interventions: Dietary Supplement: Safr'Inside supplement (Activ'Inside, SAS)
- Control group (Placebo Comparator): The Control group will take a single placebo capsule (matched to the experimental intervention in terms of colours and taste, without the active compounds saffron) twice daily (one morning and one evening after the meal).
  Interventions: Other: Plcebo

INTERVENTIONS:
Dietary Supplement: Safr'Inside supplement (Activ'Inside, SAS) — Dietary supplementation will be taken in addition to habitual diet of the patients
  Arms: Saffron extract supplementation (15mg, twice daily)
Other: Plcebo — Placebo capsule (matched to the experimental intervention in terms of colours and taste, without the active compounds saffron)
  Arms: Control group

SUMMARY:
The aim of the present study is to assess the effects of a normalised saffron extract supplementation, which is an extract of the flower Crocus sativus, on perimenopausal symptoms.

DETAILED DESCRIPTION:
After being informed about the study protocol aim and potential risks, healthy volunteer woman (walk-in outpatients) will undergo a pre-screening to determine eligibility for study entry. At the visit 1, patients who meet the pre-screening criteria will undergo a second screening to confirm their eligibility based on inclusion and exclusion criteria. After signing the inform consent form, patient who meet eligibility criteria will be randomised in a double-blind manner (participants and investigators) in a 1:1 ratio to saffron extract supplementation (15mg, twice daily) or matched placebo (twice daily) for a period of 3-months (12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Biological Female which identify themselves as Women
* Aged ≥ 40 years
* Irregular menstrual cycle for at least 3 months
* Presenting typical symptoms of perimenopause with GCS score over 20
* BMI range between 18-35 kg/m2
* Healthy woman

Exclusion Criteria:

* Less than 40 years old
* Pregnant
* Diagnosed with diseases related to reproductive system such as PCOS or endometriosis
* Taking anti-depressant medication or sleeping pills
* Taking hormonal replacement therapy (HRT)
* Taking conventional drug treatment or dietary supplementation
* Having medical history or medical/surgical event in the last 6 months, or has been treated for cancer or any other ongoing treatment for the past 3 months,
* Current and/or past history of hyper/hypotension, CVD, diabetes, autoimmune diseases, musculoskeletal disorder or endocrine or immunocompromised or neurological or psychological disorders,
* Being medicated for these conditions,
* History of allergic reactions to saffron intake,
* Decisionally challenged subjects or unable to comply to the study
* Any conditions that could contraindicates the use of saffron
* Currently smoking or ceased smoking in the past 3 months

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biologically characterised as Female
Enrollment: 104 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect on overall perimenopause clinical symptoms severity | 6-weeks, 12-weeks
  Changes in Greene Climacteric Scale (GCS) score

SECONDARY OUTCOMES:
Effect on sleep quality | 6-weeks, 12-weeks
  Changes in Pittsburg sleep quality index (PSQI) score
Effect on mood | 6-weeks, 12-weeks
  Changes in Profile of Mood State (POMS) score
Effect on quality of life | 6-weeks, 12-weeks
  Changes in Short Form Health Survey (SF-36) score
Exploratory measures | 12-weeks
  Changes in fasting plasma glucose level
Exploratory measures | 12-weeks
  Changes in gut microbiome (16S RNA Seq)
Exploratory measures | 12-weeks
  Changes in FSH levels
Exploratory measures | 12-weeks
  Changes in LH levels
Exploratory measures | 12-weeks
  Changes in TSH levels

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biochemistry, LUMHS, Jāmshoro, Sindh, Pakistan